CLINICAL TRIAL: NCT00179855
Title: Extracorporeal Photopheresis for Steroid-refractory Acute GVHD in Children and Young Adults: a Safety and Feasibility Study.
Brief Title: Extracorporeal Photopheresis for Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 0703
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Graft Versus Host Disease; Cancer; Stem Cell Transplantation
Keywords: graft versus host disease; ECP; extracorporeal photopheresis; allogeneic transplantation
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — ECP will be performed using the UVAR® XTS™ photopheresis system (Therakos). Whole blood is drawn and separated by centrifuge to collect the buffy coat (lymphocyte solution). Methoxsalen (8-MOP) is added to the blood, and the final solution of cells is passed as a film, 1mm thick, through a disposable plastic device, exposed to a UVA light source (2J/cm2/cell) and then returned to the patient.
  ECP will be performed weekly on 2 consecutive days for 4 weeks. After 4 weeks the interval will be prolonged to every 2 weeks and ECP will be stopped after maximal response has been maintained for 2 weeks. The actual study finishes at d56 but ECP may be continued beyond that (off-study) at the discretion of the physician.

SUMMARY:
The purpose of this research study is to evaluate the safety and feasibility of extracorporeal photopheresis (ECP) in the treatment of steroid-refractory acute graft-versus-host disease (GVHD) in children.

ELIGIBILITY:
Inclusion Criteria:

* Status-post allogeneic stem cell transplant (includes cord blood transplant, matched-unrelated-donor transplant and matched-related donor transplant) for any indication.
* HLA matching needs to be 4-6/6 by at least intermediate resolution for class I + II for cord blood and 5-6/6 for matched related or matched unrelated donors.
* Diagnosis of grade II-IV acute GVHD with histological confirmation of at least one organ (skin, gut, or liver) within the last 14 days. Grading of acute GVHD is per the standard Keystone criteria. Prior to enrollment, efforts should be made to rule out diagnoses that may mimic GVHD, such as drug rashes or GI infection. Patients that are being treated for acute GVHD and appear to be progressing to chronic GVHD are also eligible
* No improvement, or worsening, of acute GVHD after at least 4 days of IV methylprednisolone dosed at, at least 2.0mg/kg/day..
* Weight >25.0kg.
* Adequate venous access.

Exclusion Criteria:

* Evidence of veno-occlusive disease.
* Intubated patient.
* Patient receiving dialysis.
* Age > 30.
* Total bilirubin >15mg/dL

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2003-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and feasibility of extracorporeal photopheresis (ECP) in the treatment of steroid-refractory acute graft-versus-host disease (GVHD) in children. | To end of study
To estimate the response rate of ECP in steroid-refractory acute GVHD in children. | To end of study

SECONDARY OUTCOMES:
To evaluate the immunological mechanisms of ECP in acute GVHD. | To end of study

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, MD, Study Director — Ann & Robert H Lurie Children's Hospital of Chicago; Sonali Chaudhury, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States